CLINICAL TRIAL: NCT02940405
Title: Effect of Ketorolac Premedication on Anesthetic Efficiency of Inferior Alveolar Nerve Block, Pre-Treatment and Post-Endodontic Pain in Teeth With Irreversible Pulpitis: A Randomized Controlled Double Blinded Trial
Brief Title: Ketorolac Premedication for Anesthetic Efficiency of IANB & Postendodontic Pain in Teeth With Irreversible Pulpitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Laila Zakaria Ismail, Resident at endodontic departement , Faculty of Oral and Dental medicine ,Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CEBC-CU-2016-10-148
Record Dates: First submitted 2016-10-19; First posted 2016-10-20 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Irreversible Pulpitis
Keywords: Ketorolac Premedication; Anesthetic Efficiency; Post-Endodontic Pain; Post-operative pain; Irreversible Pulpitis; Oral premedication
MeSH Terms: conditions — Pain, Postoperative | interventions — Ketorolac Tromethamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ketorolac tromethamine (Experimental): One tablet of Ketorolac tromethamine 10-mg one hour before endodontic treatment
  Interventions: Drug: Ketorolac Tromethamine
- placebo tablet (Placebo Comparator): One tablet of a placebo one hour before endodontic treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketorolac Tromethamine — A 10 mg tablet of the medication will be given one hour before starting the root canal treatment
  Other Names: ketolac, toradol
  Arms: ketorolac tromethamine
Drug: Placebo — The placebo given as a tablet one hour before staring the root canal treatment
  Arms: placebo tablet

SUMMARY:
The aim of this study to assess effect of ketorolac premedication on the effectiveness of the inferior alveolar nerve block, pretreatment and postoperative pain in patients with symptomatic irreversible pulpitis.

DETAILED DESCRIPTION:
* Patients will be clinically and radiographically examined and their eligibility will be assessed and preoperative pain will be measured. Eligible patients will be treated in one visit.
* Patients will be randomly assigned to one of 2 groups: experimental group (taking a 10 mg tablet of ketorolac) and the control group (taking a placebo tablet). Each tablet will be taken one hour before starting treatment. The patient's pain will be assessed before local anesthetic adminstration. After 15 minutes of the initial inferior alveolar nerve block (IANB), the teeth will be examined using a cold pulp sensitivity test; in case of no or mild pain, the treatment will be initiated.
* During root canal treatment, no to mild pain response will be considered success. In case of failure, supplemental anesthesia will be administrated.
* Postoperative pain will be assessed 6, 12, 24 and 48 hours after treatment. The number of patients who will require rescue analgesic medication within the 48 hours postoperatively will be counted.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-45 years old.
2. Males or Females.
3. Mandibular Posterior teeth with symptomatic irreversible pulpitis.
4. Patients with non-contributory systemic condition.

Exclusion Criteria:

1. Patients allergic to any analgesics or antibiotics or anesthetics
2. Pregnant females
3. If analgesics have been administrated during the past 8 hours before endodontic treatment.
4. Irrestorable teeth.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-10 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Anesthetic efficiency | Intraoperative (During endodontic treatment)
  Pain during endodontic treatment will be assessed using a numerical rating scale (NRS). No or mild pain response will be considered success.

SECONDARY OUTCOMES:
Postoperative pain | At 6,12, 24, 48 hours after root canal treatment
  Postoperative pain will be measured using a numerical rating scale (NRS)
Number of patients requiring rescue analgesic. | Within 48 hours after endodontic treatment
  Number of patients requiring rescue analgesic within 48 hours after endodontic treatment

CONTACTS AND LOCATIONS:
Overall Officials: Laila Z Ismail, Postgraduate, Principal Investigator — Cairo University; Suzan AW Amin, PhD, Study Chair — Cairo University; Salsabeel M Ibrahim, Professor, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saha SG, Jain S, Dubey S, Kala S, Misuriya A, Kataria D. Effect of Oral Premedication on the Efficacy of Inferior Alveolar Nerve Block in Patients with Symptomatic Irreversible Pulpitis: A Prospective, Double-Blind, Randomized Controlled Clinical Trial. J Clin Diagn Res. 2016 Feb;10(2):ZC25-9. doi: 10.7860/JCDR/2016/16873.7195. Epub 2016 Feb 1. PMID 27042580
- [Background] Aggarwal V, Singla M, Kabi D. Comparative evaluation of effect of preoperative oral medication of ibuprofen and ketorolac on anesthetic efficacy of inferior alveolar nerve block with lidocaine in patients with irreversible pulpitis: a prospective, double-blind, randomized clinical trial. J Endod. 2010 Mar;36(3):375-8. doi: 10.1016/j.joen.2009.11.010. PMID 20171350
- [Background] Sethi P, Agarwal M, Chourasia HR, Singh MP. Effect of single dose pretreatment analgesia with three different analgesics on postoperative endodontic pain: A randomized clinical trial. J Conserv Dent. 2014 Nov;17(6):517-21. doi: 10.4103/0972-0707.144574. PMID 25506136
- [Background] Jena A, Shashirekha G. Effect of preoperative medications on the efficacy of inferior alveolar nerve block in patients with irreversible pulpitis: A placebo-controlled clinical study. J Conserv Dent. 2013 Mar;16(2):171-4. doi: 10.4103/0972-0707.108209. PMID 23716973